CLINICAL TRIAL: NCT04571749
Title: Handoffs and Transitions in Critical Care - Understanding Scalability
Acronym: HATRICC-US
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 843670; R01HL153735 (NIH)
Record Dates: First submitted 2020-07-30; First posted 2020-10-01 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Patient Handoff; Healthcare Team; Communication; Patient Safety; Intensive Care Units
Keywords: Implementation; Quality Improvement; Patient Safety; Handoffs; Intensive Care Unit; Postoperative Care
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Customized Or to ICU handoff protocol (Experimental): Tailored implementation strategies will be used in 12 ICUs to facilitate the uptake and sustained use of a customized handoff protocol to be used by clinicians at the time of patient care transition from the operating room to the intensive care unit.
  Interventions: Behavioral: Customized handoff

INTERVENTIONS:
Behavioral: Customized handoff — A customized handoff will be implemented that consists of choreographed handoffs utilizing a structured handoff tool to facilitate information exchange.

SUMMARY:
The investigators will leverage implementation science and engineering to adapt, implement, and rigorously evaluate tailored postoperative handoff protocols and implementation strategies. In doing so, the investigators will develop a vital understanding of the factors needed for successful and sustained use of evidence-based interventions in acute care. This knowledge will inform approaches to bridge the evidence-to-practice gap that prevents effective interventions from realizing the promise of improved patient outcomes in acute care settings.

DETAILED DESCRIPTION:
Surgical patients who require post-surgical critical care are usually transferred from the operating room (OR) to the intensive care unit (ICU) for ongoing care. The process of transferring the patient from the OR to the ICU is called a "handoff." Handoffs involve the transfer of patient information and transfer of patient care responsibilities from the OR team to the ICU team. Multiple studies suggest that these handoffs can expose patients to preventable harm, which can be avoided with standardization of the handoff. The Handoffs and Transitions in Critical Care (HATRICC; IRB #819726) study, started in 2014, developed and implemented a standardized OR to ICU handoff process in two Penn surgical ICUs (SICUs) that did not have a standardized handoff process.

Four clinicians (surgeon, anesthetist, ICU provider, and ICU nurse) from two teams (surgical and intensive care) usually take part in handoff communication. During the HATRICC study, the investigators evaluated handoff communication between the OR and ICU teams before and after implementation of the new standardized handoff process (the "HATRICC process") in multiple ways, using observations, interviews, focus groups, and surveys. The investigators demonstrated a 20% improvement in information exchange after implementation of the HATRICC standardized handoff process, a process tailored to meet the needs of the different clinicians participating in OR to ICU handoffs.

Prior studies have indicated short-term success in standardizing OR to ICU handoffs, but sustainability of these improvement interventions has been less well studied. Two studies have demonstrated sustained or improved information exchange following the institution of structured OR to ICU handoff processes, but the factors influencing sustainability remain to be elucidated.

The aims of this study are to:

1. Ascertain determinants of OR-to-ICU handoff protocol adoption and use in 12 adult and pediatric ICUs in five health systems.
2. Adapt handoff protocols using engineering approaches and select tailored implementation strategies with implementation mapping.
3. Test the effectiveness of tailored, multifaceted, multilevel implementation strategies.
4. Design and create a digital toolkit for other ICUs to identify implementation determinants, customize OR-to-ICU handoff protocol, and select appropriate implementation strategies.

ELIGIBILITY:
Inclusion Criteria for Clinicians:

* Age ≥ 18 years
* Cares for patients at any point in the surgical continuum of care, including pre-operative, intra-operative, or post-operative care, OR has administrative responsibilities relevant to patient care at the study hospitals
* Fluency in English

Inclusion Criteria for Patients:

• Patient admitted for inpatient care at the study hospitals and experiences a post-operative handoff from the operating room to the intensive care unit.

Exclusion Criteria for Clinicians:

• Being a member of research staff

Exclusion Criteria for Patients:

• (none)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2021-04-11 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to standardized handoff intervention (Fidelity) measured by number of handoff steps followed. | This outcome will be measured at monthly intervals starting Year 1, Quarter 2 and continuing until the end of Year 5.
  Fidelity is defined as adherence to the standardized handoff intervention. Fidelity is a count of handoff steps followed, with scores ranging from 0 to 10. Fidelity will be measured by trained site-based observers. Field notes by trained observers will inform the interpretation of fidelity. Units of analysis: patient level (handoff level), ICU level.
New-onset organ failure | This outcome will be measured at monthly intervals starting Year 1, Quarter 2 and continuing until the end of Year5
  Per-protocol handoffs enable clinicians to follow expected care practices and to anticipate and avoid postoperative deterioration.

SECONDARY OUTCOMES:
Perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory (Acceptability) | Baseline (Year 1); within 2months of implementation; within 2 months of beginning sustainment
  Acceptability is defined as "the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory." (Proctor et al, Adm Policy Ment Health (2011) 38:65-76). Acceptability will be measured using the Acceptability of Intervention Measure (AIM) developed by Weiner et al (Implement Sci. 2017;12(1):108; see Appendix). Interview and focus group transcripts and field notes will be analyzed to develop a more nuanced understanding of acceptability. Unit of analysis: individual (employed staff)
Perceived fit, relevance, or compatibility of the innovation in a practice setting or to address a particular issue (Appropriateness), measured by the Intervention Appropriateness Measure | Baseline (Year 1); within 2months of implementation; within 2 months of beginning sustainment
  Appropriateness is defined as "the perceived fit, relevance, or compatibility of the innovation or evidence based practice for a given practice setting, provider, or consumer; and/or perceived fit of the innovation to address a particular issue or problem." (Proctor et al, Adm Policy Ment Health (2011) 38:65-76). Appropriateness will be measured using the Intervention Appropriateness Measure (IAM) developed by Weiner et al (Implement Sci. 2017;12(1):108; see Appendix). Interview and focus group transcripts and field notes will be analyzed to develop a more nuanced understanding of appropriateness. Unit of analysis: individual (employed staff)
Feasibility of treatment or innovation to be carried out in a practice setting, measured using the Feasibility of Intervention Measure. | Baseline (Year 1); within 2months of implementation; within 2 months of beginning sustainment
  Feasibility is defined as "the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting." (Proctor et al, Adm Policy Ment Health (2011) 38:65-76). Feasibility will be measured using the Feasibility of Intervention Measure (FIM) developed by Weiner et al (Implement Sci. 2017;12(1):108; see Appendix). Interview and focus group transcripts and field notes will be analyzed to develop a more nuanced understanding of feasibility. Unit of analysis: individual (employed staff)
Fidelity over time (Sustainment) | This outcome will be measured at monthly intervals starting 2 years after implementation, up to 5 years.
  Sustainment is defined as fidelity over time. We define the sustainment phase as starting two years after implementation. Units of analysis: patient level (handoff level), ICU level.
Monetary and non-monetary costs measured using the line item classification system | This outcome will be measured within 2 months of implementation; within2 months of beginning sustainment
  We will conduct a retrospective cost analysis as described by Hoeft et al (Implementation Science 2019;14(1):37). We will use the line item classification system, in which accounting principles are used to calculate costs, and will attempt to include both monetary costs and non-monetary costs (e.g., opportunity costs). Activities undertaken only for research (e.g., interviews and focus groups) will not be included in this analysis. Field notes will be the primary data source for this outcome. Unit of analysis: ICU level.
Teamwork (effectiveness) measured using the Team Emergency Assessment Measure. | This outcome will be measured at quarterly intervals starting Year 1, Quarter 2 and continuing until the end of Year 5
  Teamwork will be measured using a validated instrument, the Team Emergency Assessment Measure (TEAM) (Cooper et al, Resuscitation 2010;81(4):446-452). Unit of analysis: handoff team.
Clinician satisfaction measured at the individual level. | This outcome will be measured annually from Years 1 to 5.
  Clinician satisfaction will be measured using a non-validated instrument adapted from the parent HATRICC study (see Appendix). Unit of analysis: individual.
Workload measured using the NASA Task Load Index. | This outcome will be measured at quarterly intervals starting Year 1, Quarter 2 and continuing until the end of Year 5.
  Workload is a measure of effectiveness and will be measured using the validated NASA Task Load Index.
Completeness of information exchange (Information Omissions) measured using a structured observation form. | This outcome will be measured at monthly intervals starting Year 1, Quarter 2 and continuing until the end of Year5
  Information omissions is a measure of the completeness of information exchange. It will be measured at the same time as fidelity using a structured observation form (see Appendix). Unit of analysis: patient level (handoff level).
Weighted average of the reliability-adjusted observed-to-expected ratios for component indicators of adverse events | This outcome will be measured at quarterly intervals starting Year 1, Quarter 2 and continuing until the end of Year 5.
  This is a composite measure defined by AHRQ as "the weighted average of the reliability-adjusted observed-to-expected ratios (indirect standardization of the smoothed rates) for the following component indicators: PSI 03 Pressure Ulcer Rate; PSI 06 Iatrogenic Pneumothorax Rate; PSI 07 Central Venous Catheter-Related Blood Stream Infection Rate; PSI 08 Postoperative Hip Fracture Rate; PSI 09 Perioperative Hemorrhage or Hematoma Rate; PSI 10 Postoperative Physiologic and Metabolic Derangement Rate; PSI 11 Postoperative Respiratory Failure Rate; PSI 12 Perioperative Pulmonary Embolism or Deep Vein Thrombosis Rate; PSI 13 Postoperative Sepsis Rate; PSI 14 Postoperative Wound Dehiscence Rate; PSI 15 Accidental Puncture or Laceration Rate." We note that some of the components of this measure overlap with our primary effectiveness outcome. Unit of analysis: ICU-level.
AHRQ PSI 9: Perioperative hemorrhage or hematoma rate(effectiveness) | This outcome will be measured at monthly intervals starting Year 1, Quarter 2 and continuing until the end of Year 5
  This measure is one of the five components of the co-primary outcome of new-onset organ failure. It is defined by AHRQ as "perioperative hemorrhage or hematoma cases with control of perioperative hemorrhage, drainage of hematoma, or a miscellaneous hemorrhage- or hematoma-related procedure following surgery per 1,000 surgical discharges." AHRQ collects this information for patients aged 18 and older, but we will collect this outcome for pediatric patients in the two pediatric ICUs. Unit of analysis: ICU-level.
AHRQ PSI 10: Postoperative physiologic or metabolic derangement rate (effectiveness) | This outcome will be measured at monthly intervals starting Year 1, Quarter 2 and continuing until the end of Year 5.
  This measure is one of the five components of the co-primary outcome of new-onset organ failure. It is defined by AHRQ as "postoperative acute renal failure (secondary diagnosis) with dialysis per 1,000 elective surgical discharges." AHRQ collects this information for patients aged 18 and older, but we will collect this outcome for pediatric patients in the two pediatric ICUs. Unit of analysis: ICU-level.
AHRQ PSI 11: Postoperative respiratory failure rate (effectiveness) | This outcome will be measured at monthly intervals starting Year 1, Quarter 2 and continuing until the end of Year 5
  This measure is one of the five components of the co-primary outcome of new-onset organ failure. It is defined by AHRQ as "postoperative respiratory failure (secondary diagnosis), prolonged mechanical ventilation, or reintubation cases per 1,000 elective surgical discharges." AHRQ collects this information for patients aged 18 and older, but we will collect this outcome for pediatric patients in the two pediatric ICUs. Unit of analysis: ICU-level.
AHRQ PSI 12: Perioperative pulmonary embolism or DVT rate (effectiveness) | This outcome will be measured at monthly intervals starting Year 1, Quarter 2 and continuing until the end of Year 5
  This measure is one of the five components of the co-primary outcome of new-onset organ failure. It is defined by AHRQ as "perioperative pulmonary embolism or deep vein thrombosis (secondary diagnosis) per 1,000 surgical discharges." AHRQ collects this information for patients aged 18 and older, but we will collect this outcome for pediatric patients in the two pediatric ICUs. Unit of analysis: ICU-level.
AHRQ PSI 13: Post operative sepsis rate (effectiveness) | This outcome will be measured at monthly intervals starting Year 1, Quarter 2 and continuing until the end of Year 5
  This measure is one of the five components of the co-primary outcome of new-onset organ failure. It is defined by AHRQ as "postoperative sepsis cases (secondary diagnosis) per 1,000 elective surgical discharges." AHRQ collects this information for patients aged 18 and older, but we will collect this outcome for pediatric patients in the two pediatric ICUs. Unit of analysis: ICU-level.
Professionalism of handoff team during handoff. | At quarterly intervals starting Year 1, Quarter 2 and continuing until the end of Year 5.
  Professionalism will be characterized qualitatively using field notes from trained observers. Unit of analysis: handoff team.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan B Lane-Fall, MD, MSHP, Principal Investigator — University of Pennsylvania
Locations (5):
- United States (5):
  - Johns Hopkins, Baltimore, Maryland
  - Cooper Health, Camden, New Jersey
  - Temple Health, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lane-Fall MB, Christakos A, Russell GC, Hose BZ, Dauer ED, Greilich PE, Hong Mershon B, Potestio CP, Pukenas EW, Kimberly JR, Stephens-Shields AJ, Trotta RL, Beidas RS, Bass EJ. Handoffs and transitions in critical care-understanding scalability: study protocol for a multicenter stepped wedge type 2 hybrid effectiveness-implementation trial. Implement Sci. 2021 Jun 15;16(1):63. doi: 10.1186/s13012-021-01131-1. PMID 34130725
- See also: HATRICC Website — http://www.hatricc.us/